CLINICAL TRIAL: NCT07023237
Title: Three-Dimensional Guidance for Pulmonary Vein Isolation in Patients With Paroxysmal Atrial Fibrillation: A Study on Efficacy and Safety
Brief Title: 3D-Guided Pulsed Field Ablation for Paroxysmal AF
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PFA
Record Dates: First submitted 2025-04-29; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation (AF); Pulsed Field Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pulsed field ablation — Pulsed electric fields refer to the generation of high-voltage electric fields with pulse widths ranging from milliseconds to microseconds or even nanoseconds. These fields release extremely high energy in a very short time, creating a large number of irreversible micropores in the cell membrane and even intracellular organelles such as the endoplasmic reticulum, mitochondria, and nucleus. This ultimately leads to apoptosis of the diseased cells, achieving the desired therapeutic effect.
  By inserting a pulsed ablation catheter into the patient's body and reaching the target lesion, the pulsed energy is delivered to the ablation catheter via a cardiac pulsed field ablation device, thereby achieving the therapeutic goal of pulsed field ablation.

SUMMARY:
Atrial fibrillation (AF) is a common arrhythmia, especially in the elderly, and can lead to severe complications like stroke and heart failure. In China, AF affects approximately 20 million adults, and its prevalence is expected to rise due to aging [1, 2]. Catheter ablation has become a first-line treatment for AF, with pulsed field ablation (PFA) gaining attention due to its tissue selectivity and non-thermal ablation properties [3-8]. PFA uses high-voltage electric fields to create cell membrane perforations, leading to permanent tissue damage and effective arrhythmia treatment [6-8].

Recent studies have shown that PFA is highly effective and safe. For example, the EU-PORIA study reported a 99.96% pulmonary vein isolation (PVI) rate with a 3.6% complication rate [9, 10], while the ADVENT study demonstrated similar efficacy to thermal ablation but with shorter procedure times [12]. However, current PFA systems often lack integration with 3D mapping systems, limiting their application in complex cases and increasing reliance on fluoroscopy [13, 14].

In China, domestic PFA technology is rapidly evolving, with a focus on expanding indications and integrating 3D techniques [19, 20]. The investigators have conducted preliminary studies on the feasibility and safety of domestic PFA in persistent AF treatment [21]. To further advance PFA, larger-scale clinical studies are needed to optimize procedural workflows and reduce complications.

This study aims to enroll 430 participants through a single-center, single-arm approach. By following up for one year, the investigators will optimize the PFA procedure under 3D guidance to enhance success rates and safety. This will support the clinical promotion of PFA technology and provide valuable data for the development of domestic PFA devices.

ELIGIBILITY:
**Inclusion Criteria:**

1. Aged 18 years or older, regardless of gender.
2. Patients with paroxysmal atrial fibrillation scheduled for catheter ablation.
3. Willing and able to comply with all follow-up requirements and agree to participate in this study.

**Exclusion Criteria:**

1. Previous left atrial catheter ablation.
2. Left ventricular ejection fraction (LVEF) < 35%.
3. Left atrial diameter (assessed by echocardiography) > 55 mm.
4. Presence of definite thrombus in the left atrium or any other cardiac chamber detected before surgery.
5. Patients with New York Heart Association (NYHA) functional class III-IV heart failure.
6. Patients with second-degree (Type II) or third-degree atrioventricular block.
7. Significant congenital heart defects (e.g., atrial septal defect or severe pulmonary vein stenosis, but not including patent foramen ovale).
8. Patients with prosthetic heart valves.
9. Patients with implanted cardiac pacemakers or implantable cardioverter-defibrillators (ICDs).
10. Patients diagnosed with hypertrophic cardiomyopathy, chronic obstructive pulmonary disease, or myxoma.
11. Patients with known symptomatic carotid artery stenosis before surgery.
12. Patients with untreated or uncontrolled hyperthyroidism or hypothyroidism.
13. Patients with systemic active infections.
14. Patients with significant bleeding tendencies or those undergoing hemodialysis for renal failure.
15. Patients who have experienced a myocardial infarction or undergone any cardiac intervention/open-heart surgery within the past 3 months.
16. Patients who have had a stroke or transient ischemic attack within the past 6 months.
17. Patients with significant contraindications to interventional procedures, as determined by the investigator, who are unable to undergo ablation surgery.
18. Pregnant or breastfeeding women, or those planning to conceive during the study period.
19. Patients who have participated in other drug or medical device clinical trials within the past 3 months.
20. Patients whom the investigator deems unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with paroxysmal atrial fibrillation scheduled for radiofrequency ablation.
Sampling Method: Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
12-Month Postoperative Treatment Success Rate | 12 months
  Definition of 12-Month Postoperative Treatment Success: No recurrence of atrial arrhythmias (atrial fibrillation, atrial tachycardia, or unexplained atrial flutter) lasting ≥30 seconds from 3 months to 12 months postoperatively, and no occurrence of any of the following failure modes: immediate procedural failure, repeat ablation failure (more than 1 repeat ablation during the blanking period, or any repeat ablation outside the blanking period), antiarrhythmic drug (AAD) failure (use of new Class I/III AADs for treatment of atrial fibrillation, atrial tachycardia, or unexplained atrial flutter, or increased dosage of previously failed Class I/III AADs), persistent atrial fibrillation/atrial tachycardia/atrial flutter documented by standard 12-lead ECG, or failure of electrical cardioversion.
  Calculation: 12-Month Postoperative Treatment Success Rate = (Number of patients with treatment success at 12 months / Total number of patients completing 12-month follow-up) × 100%

SECONDARY OUTCOMES:
Immediate Procedural Success Rate | immediately after procedure
  Definition of Immediate Procedural Success: Achievement of complete pulmonary vein isolation and superior vena cava isolation after ablation.
  Calculation: Immediate Procedural Success Rate = (Number of patients with immediate procedural success / Total number of patients undergoing the procedure) × 100%
Success Rate of No Recurrence of Atrial Arrhythmias (≥30 seconds) Without Class I/III AADs from 3 Months to 12 Months Postoperatively | 12 months

IPD SHARING:
Plan to Share IPD: No